CLINICAL TRIAL: NCT07367178
Title: Phase II Study to Improve Sacituzumab Govitecan Tolerance With Atropine in Patients With Advanced Triple-Negative and Hormone Receptor-Positive/HER2-Negative Breast Cancer
Brief Title: Study of Sacituzumab Govitecan With Atropine to Improve Tolerability in Advanced TNBC and HR+/HER2- Breast Cancer
Acronym: SATROPIN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDOPP824; 2025-524109-33-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Advanced HR+/HER2- Breast Cancer; Advanced Triple-Negative Breast Cancer
Keywords: Advanced TNBC; Sacituzumab govitecan; Atropine; Tolerance; Advanced HR+/HER2-; Prophylaxis; SATROPIN
MeSH Terms: conditions — Breast Neoplasms | interventions — sacituzumab govitecan; Atropine; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Intervention Model Description: International, multicenter, open-label, single-arm, phase II clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab govitecan + Atropine + G-CSF (Experimental): After having confirmed eligibility and enrollment into the clinical trial, participants will receive sacituzumab govitecan at a dose of 10 mg/kg body weight, administered via intravenous (IV) infusion on Day 1 and Day 8 of each 21-day cycle. Subcutaneous atropine sulfate at a dose of 0.5 mg will be given as premedication prior to each sacituzumab govitecan infusion during the first two treatment cycles. Continuation of atropine beyond Cycle 2 will be at the discretion of the Investigator. Participants will be treated until unacceptable toxicity, disease progression, withdrawal of consent, death, or study termination, whichever occurs first. To improve hematologic tolerability, G-CSF will be used as a supportive medication during the first 2 cycles of sacituzumab govitecan. The use of G-CSF beyond the second cycle will be at the discretion of the Investigator.
  Interventions: Drug: Sacituzumab Govitecan (SG); Drug: Atropine; Drug: G-CSF (Granulocyte colony-stimulating factor)

INTERVENTIONS:
Drug: Sacituzumab Govitecan (SG) — Participants will receive sacituzumab govitecan at a dose of 10 mg/kg body weight, administered via intravenous (IV) infusion on Day 1 and Day 8 of each 21-day cycle until unacceptable toxicity, disease progression, death, discontinuation from the Study treatment for any other reason or End of the Study (EoS), whichever occurs first.
  Other Names: Trodelvy
Drug: Atropine — Participants will receive atropine at a dose of 0.5 mg as premedication 10 minutes before prior to each sacituzumab govitecan infusion during the first two treatment cycles. Continuation of atropine beyond Cycle 2 will be at the discretion of the Investigator.
Drug: G-CSF (Granulocyte colony-stimulating factor) — All participants will receive 0.5MU/kg/day of G-CSF, according to the participant's weight, which will be administered subcutaneously (SC), once a day during two consecutive days, 48 hours after administration of sacituzumab govitecan (D3, D4 and D10, D11) during the first two cycles. The use of G-CSF beyond the second treatment cycle will be at the discretion of the Investigator.
  Other Names: Filgrastim; non-PEGylated G-CSF

SUMMARY:
The SATROPIN study is an international, multicenter, open-label, single-arm, phase II clinical trial to assess whether the use of prophylactic administration of atropine may prevent diarrhea in participants with unresectable locally advanced or metastatic triple-negative breast cancer (TNBC) or hormone receptor-positive/HER2-negative (HR(+)/HER2-) treated with sacituzumab govitecan.

DETAILED DESCRIPTION:
After signing the informed consent form (ICF) and confirmation of eligibility, participants with mTNBC or mHR(+)/HER2(-) breast cancer will receive sacituzumab govitecan administered as intravenous infusion (IV) at dose of 10 mg/kg on D1 and D8 of each 21-day cycle until unacceptable toxicity, disease progression, withdrawal of consent, death, or study termination, whichever occurs first. Atropine will be administered 0.5 mg SC as premedication 10 minutes before each infusion of sacituzumab govitecan on D1 and D8 of each 21-day cycle during the first two treatment cycles (consider extending to the next cycles at the discretion of the physician). To improve hematologic tolerability, G-CSF will be used as a supportive medication during the first 2 cycles of sacituzumab govitecan. The use of G-CSF beyond the second treatment cycle will be at the discretion of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Participant, or legal representative (if applicable), must be capable of understanding the purpose of the Study and have signed a written informed consent form (ICF) prior to beginning specific protocol procedures.
2. Female or male participants ≥ 18 years of age at the time of signing ICF.
3. ECOG performance status of 0 or 1.
4. Minimum life expectancy of ≥ 12 weeks at screening.
5. Unresectable locally advanced or metastatic disease documented by computerized tomography (CT) scan or magnetic resonance imaging (MRI) that is not amenable to curative therapy.
6. For TNBC participants only:

   i. Histologically confirmed TNBC of the most recent available sample per American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) 2018 criteria on the most recently analyzed biopsy. TNBC status is defined as <1% expression for estrogen receptor (ER) and progesterone receptor (PgR) and negative for human epidermal growth factor receptor 2 (HER2) (0-1+ by immunohistochemistry [IHC] or 2+ and negative by in situ hybridization [ISH] test).
7. For HR(+)/HER2(-) breast cancer participants only:

   i. Histologically confirmed HR(+)/HER2(-) breast cancer of the most recent available sample per ASCO/CAP 2018 criteria on the most recently analyzed biopsy. HR(+)/HER2(-) status is defined as ≥1% expression for ER and/or PgR and negative for HER2 (0-1+ by IHC or 2+ and negative by ISH test).

   ii. Disease progression to at least one prior endocrine therapy for advanced disease.

   iii. Disease progression to previous CDK4/6i-based therapy in any setting. For participants who received CDK4/6i in the adjuvant setting, a minimum of one year of treatment and a disease-free interval (DFI) of ≤12 months are required.

   Note: For participants with ER-low positive tumor (defined as ER expression between 1% and 10%) previous therapy with CDK4/6 inhibitors and/or endocrine therapy is permitted but not required.
8. Disease progression to no more than two prior standard of care chemotherapy-based regimens for advanced disease (prior ADC will count as a chemotherapy-based regimen).

   Note: Earlier adjuvant or neoadjuvant therapy for early breast cancer will be considered as one of the required prior regimens if the development of unresectable locally advanced or metastatic disease occurred within a 12-month period after treatment completion.
9. Prior treatment with a trophoblast cell-surface antigen 2 (TROP2) ADC and/or topoisomerase I inhibitor or an ADC containing a topoisomerase I inhibitor is only allowed in the (neo)adjuvant setting if the development of unresectable locally advanced or metastatic disease occurred at least 12 months after treatment completion.
10. Measurable or non-measurable, but evaluable disease, as per RECIST v.1.1.
11. Participants must have adequate bone marrow, liver, and renal function:

    i. Adequate hematologic counts without transfusion or growth factor support within two weeks before of study drug initiation (hemoglobin ≥ 9 g/dL, ANC ≥ 1500/mm3, and platelets ≥ 100,000/ μL).

    ii. Adequate renal and hepatic function (creatinine clearance of ≥ 60 ml/min, may be calculated using Cockcroft-Gault equation; bilirubin ≤ 1.5 x ULN and AST/ALT ≤ 3.0 x ULN or 5 x ULN if known liver metastases).

    Note: Participants with a known or genetically confirmed Gilbert's syndrome (based on UGT1A1 polymorphism testing) may be enrolled provided that total bilirubin is <1.5 × ULN. The diagnosis of Gilbert's syndrome must be recorded in the patient's medical history, and if UGT1A1 status is available, the type of mutation should also be documented.
12. Participants must be willing to provide the most recent archival tumor tissue sample (from the primary breast tumor or a metastatic site) at baseline, as well as biological samples (blood and stool) at the established time points.
13. Resolution of all acute toxic effects of prior anticancer therapy to grade ≤1 as determined by the US National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 6.0 (v.6.0) (except for alopecia or other toxicities not considered a safety risk for the participant at investigator's discretion).
14. Women of childbearing potential who are sexually active with a non-sterilized male partner must have a negative serum pregnancy test within 14 days before Study treatment initiation. In addition, they must agree to use one highly effective method of birth control from the time of screening until six months after the last dose of Study treatment. Female participants must refrain from egg cell donation and breastfeeding during this same period.
15. Male participants who are sexually active with a female partner of childbearing potential must be surgically sterile or using an acceptable method of contraception from the time of screening until three months after the last administration of Study treatment. Male participants must not donate or bank sperm during this same period.
16. Participants must be accessible for treatment and follow-up.

Exclusion Criteria:

1. Participation in another clinical trial, interventional or observational, until the Study's safety visit.

   Note: Participation in retrospective studies or data analysis is allowed.
2. Known leptomeningeal disease or active uncontrolled or symptomatic central nervous system (CNS) metastases as indicated by clinical symptoms, and/or progressive growth are excluded.

   Note: Participants with a history of CNS metastases are eligible if they have been previously treated with local therapy, are clinically stable, and off anticonvulsants and steroids for at least 14 days before the first dose of Study treatment.
3. Have a concurrent malignancy or malignancy within three years of Study enrollment with the exception of carcinoma in situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin that has been previously treated with curative intent. For other cancers considered to have a low risk of recurrence, discussion with the Sponsor's Medical Monitor is required.
4. Known allergy or hypersensitivity reaction to any investigational medicinal product(s) (IMP[s]) or its (their) incorporated substances.
5. Participants at risk of urinary retention (e.g.,those with prostatic hypertrophy), prior history of glaucoma, both open and closed angle, and previous diagnosis of myasthenia gravis, conditions in which atropine is contraindicated.
6. Requirement for ongoing therapy with any prohibited medications listed in the protocol.
7. Have received prior radiotherapy within two weeks before the first dose of Study treatment (four weeks in case of radiation therapy of the central nervous system). Participants must have recovered from all radiation-related toxicities, not require steroids.
8. Major surgical procedure or significant traumatic injury within 14 days before the first dose of Study treatment or anticipation of need for major surgery within the course of the Study treatment.
9. Known history of unstable angina, myocardial infarction, or cardiac heart failure present within six months of study initiation or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy or history of QT interval prolongation.
10. Clinically significant active pulmonary compromise at screening (e.g., ongoing infection, uncontrolled COPD/asthma exacerbation).

    Note: Participants with stable chronic lung diseases (e.g., controlled COPD, asthma, bronchiectasis, post-COVID fibrosis) may be enrolled but atropine should be used with caution and participants should be monitored for respiratory complications.
11. Known history of clinically significant bleeding, thrombosis, intestinal obstruction, or gastrointestinal perforation within six months of study initiation.
12. Documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or a preexisting chronic condition resulting in baseline grade ≥1 diarrhea).
13. Any other serious medical condition and/or abnormality in clinical laboratory tests that, in the Investigator's judgment, precludes the participant's safe participation in and completion of the Study.
14. Current known infection with hepatitis B virus (HBV), or hepatitis C virus (HCV). Participants with past HBV infection or resolved HBV infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV DNA test) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
15. Active primary immunodeficiency, known human immunodeficiency virus (HIV) infection.

    i. Note: Participants with HIV on antiretroviral therapy (ART) with well-controlled HIV infection/disease are allowed.

    ii. Participants on ART must have a CD4+ T-cell count ≥ 350 cells/mm3 at time of screening.

    iii. Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 copies/mL or the lower limit of qualification (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks prior to screening.

    iv. Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks prior to Study entry.

    v. The combination of the ART regimen must not contain any medications that may interfere with SN-38 metabolism (such as CYP3A4 inhibitors or inducers as raltegravir, nevirapine, or atazanavir).
16. Other active uncontrolled infection at the time of enrollment.
17. Receipt of live or attenuated vaccine within 30 days prior to the first dose of Study treatment.
18. Pregnant or lactating women or participants not willing to apply highly effective contraception as defined in the protocol.
19. Treatment with approved or investigational cancer therapy within 14 days prior to initiation of Study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To assess the incidence and severity of diarrhea during the first two treatment cycles | Baseline up to end of 2nd cycle (day 42)
  Incidence of grade ≥2 diarrhea during the first two treatment cycles as assessed by the Investigator, with severity determined by the NCI-CTCAE v.6.0.

SECONDARY OUTCOMES:
To assess the incidence and severity of constipation during the first two treatment cycles | Baseline up to end of 2nd cycle (day 42)
  Incidence of all grades constipation during the first two treatment cycles, as assessed by the Investigator, with severity determined by the NCI-CTCAE v.6.0.
To determine the overall safety profile during the first two treatment cycles and the extended follow-up. | Until EoS (9 months after last participant is included in the Study unless premature termination of the Study)
  Overall safety profile according to the NCI-CTCAE v.6.0 during the first two treatment cycles and the extended follow-up
To evaluate the incidence and severity of diarrhea during the first two treatment cycles versus extended follow-up. | Until EoS (9 months after last participant is included in the Study unless premature termination of the Study)
  Incidence of all grades diarrhea during the first two treatment cycles and during the extended follow-up, as assessed by the Investigator, with severity determined by NCI-CTCAE v.6.0.
To evaluate the incidence and severity of constipation during the first two treatment cycles versus extended follow-up. | Until EoS (9 months after last participant is included in the Study unless premature termination of the Study)
  Incidence of all grades constipation during the first two treatment cycles and during the extended follow-up, as assessed by the Investigator, with severity determined by NCI-CTCAE v.6.0.
To assess the dose reduction rate. | Until EoS (9 months after last participant is included in the Study unless premature termination of the Study)
  Dose reduction rate, defined as the proportion of participants with dose reduction due to toxicity relative to the number of participants in the analysis set.
To evaluate the dose interruption rate. | Until EoS (9 months after last participant is included in the Study unless premature termination of the Study)
  Dose interruption rate, defined as the proportion of participants with dose interruption due to toxicity relative to the number of participants in the analysis set.
To analyze the discontinuation rate. | Until EoS (9 months after last participant is included in the Study unless premature termination of the Study)
  Discontinuation rate, defined as the proportion of participants who discontinued Study treatment to any cause relative to the number of participants in the analysis set.
To assess real-world progression-free survival (rwPFS). | Until EoS (9 months after last participant is included in the Study unless premature termination of the Study)
  rwPFS, defined as the time between start of treatment to date of disease progression or death documented in participant medical charts, whichever date came first.
To evaluate the time to treatment failure (TTF). | Until EoS (9 months after last participant is included in the Study unless premature termination of the Study)
  TTF, defined as the time from the start of treatment to its discontinuation for any reason, including disease progression, treatment-related toxicity, participant withdrawal, or death.
To determine the time to treatment failure due to toxicity (TTF-Toxicity). | Until EoS (9 months after last participant is included in the Study unless premature termination of the Study)
  TTF-Toxicity, defined as the time from the start of treatment to its discontinuation especially due to treatment-related adverse events (TEAEs). It excludes discontinuation for other reasons such as disease progression, participant withdrawal, or death unrelated to toxicity.
To assess overall survival (OS). | Until EoS (9 months after last participant is included in the Study unless premature termination of the Study)
  OS, defined as the period from treatment initiation to death from any cause, as determined locally by the Investigator.

IPD SHARING:
Plan to Share IPD: Yes
Data collected within this study will be made available to researchers after contacting the corresponding author and upon revision and approval based on scientific merit by the trial management group (which includes a qualified statistician) of a detailed proposal for their use. The data required for the approved, specified purposes and the trial protocol will be provided after the completion of a data-sharing agreement that will be set up by the study sponsor. All data provided are anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. Data Sharing should begin 1 month after publication of study main results and ending 5 years after article publication. Estimate timeframe for response will be within 30 days.